CLINICAL TRIAL: NCT06027242
Title: Oral Supplementation of Glutamine on Gastric Cancer Patients After Gastrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Jin-Ming Wu, Clinical Associate Professor & PhD, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202207099RINA
Record Dates: First submitted 2023-08-17; First posted 2023-09-07 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer; Immunonutrition; Gastrostomy
Keywords: Gastric cancer; Gastrectomy; sarcopenia
MeSH Terms: conditions — Stomach Neoplasms; Sarcopenia | interventions — Glutamine; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without oral glutamine supplementation (Placebo Comparator): 15 g Maltodextrin for 28 days after surgery with tolerable oral intake or enteral feeding
  Interventions: Dietary Supplement: Maltodextrin
- With oral glutamine supplementation (Active Comparator): 10 g glutamine +5 g Maltodextrin for 28 days after surgery with tolerable oral intake or enteral feeding
  Interventions: Dietary Supplement: oral glutamine; Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: oral glutamine — 10 g glutamine +5 g Maltodextrin for 28 days after surgery with tolerable oral intake or enteral feeding
  Arms: With oral glutamine supplementation
Dietary Supplement: Maltodextrin — Maltodextrin

SUMMARY:
Glutamine has the potentials of immunomodulation and adjustment of protein metabolism. The primary objective of this study is to evaluate the efficacy of glutamine on sarcopenia in gastric adenocarcinoma patients undergoing gastrectomy. The secondary endpoints, including the physical activity, weight loss, and nutritional profiles, will be evaluated among these patients.

DETAILED DESCRIPTION:
This will be a double-blind, randomized, and placebo-controlled study. At least 80 evaluable patients who are scheduled for gastrectomy for gastric adenocarcinoma cancer will be randomly assigned to the control or treatment group. Each group will have at least 40 patients. The CT scan will be evaluated before surgery and on postoperative day (POD) 90. Moreover, the patient will wear the smart watch to record daily walking steps. Laboratory data will be check before gastrectomy and on POD 90.

ELIGIBILITY:
Inclusion Criteria:

* adult gastric cancer receiving gastrectomy

Exclusion Criteria:

* Hepatic insufficiency
* Renal insufficiency
* can not tolerate oral or enteral feeding 7 days after gastrectomy
* can not receive computed tomograph
* can not waer the wearable devices

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Change of area of psoas muscle | 84 days after gastrectomy
  area od psoas muscle on the CT scan

SECONDARY OUTCOMES:
Walking steps | 28,56, and 84 days after gastrectomy
  the average daily walking steps recorded by the wearable devices
body weight | 84 days after gastrectomy
  body weight
Change of serum albumin value | 84 days after gastrectomy
Change in white blood cells counts | 84 days after gastrectomy
Change in lymphocyte cells counts | 84 days after gastrectomy
Change of serum pre-albumin value | 84 days after gastrectomy

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Ming Wu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT06027242/Prot_SAP_000.pdf